CLINICAL TRIAL: NCT05415566
Title: The Effect of Therapeutic Play Applied by Using Toy Nebulizer and Toy Mask on Child's Fear and Anxiety Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ayşe Kahraman, associate professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21116
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Therapeutic Play; Anxiety; Fear
Keywords: Toy Mask; Toy Nebulizer; Child; Nurse
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The population of the randomized controlled experimental study was composed of children aged 3-8 years who applied to the pediatric emergency department due to respiratory system disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Treatment Group (No Intervention): Inhaler treatment was applied according to the routine procedure in the emergency department.
- Therapeutic Play Group (Experimental): Inhaler treatment was applied according to the "Therapeutic Play Guide" prepared by the researcher.
  Interventions: Combination Product: toy nebulizer and toy mask

INTERVENTIONS:
Combination Product: toy nebulizer and toy mask — The treatment was administered using therapeutic play.
  Arms: Therapeutic Play Group

SUMMARY:
In this study, it was aimed to examine the effect of therapeutic play applied with a toy nebulizer and toy mask before inhaler treatment on children's fear and anxiety.

It is the hypothesis of the study that the therapeutic play applied by using a toy mask and a toy nebulizer before inhaler treatment in children will reduce the child's fear and anxiety.

DETAILED DESCRIPTION:
Acute diseases constitute the majority of applications made to pediatric emergency services. Inhaled drugs are frequently used in the treatment of childhood acute respiratory system diseases. Nebulizers are the preferred method of administering inhaled drugs. Medical procedures are one of the biggest fears of children, making it difficult to use nebulizers correctly and effectively. The negative reaction of the child to the mask and nebulizer during inhaler treatment causes incorrect inhalation patterns, reducing the safety and effectiveness of the treatment. This causes difficulties in relieving symptoms, increased hospital admission and hospitalization time, more treatment costs, and even negative consequences such as increased morbidity.

Reducing the fear and anxiety seen in children due to the hospital environment and illness is important in terms of children's acceptance of the treatment process. One of the methods used for this purpose is therapeutic play. Pediatric nurses should fulfill their nursing roles and responsibilities by including therapeutic play in their care processes.

ELIGIBILITY:
Inclusion Criteria:

1. Parent and child volunteering to participate in the study,
2. The child is between the ages of 3-8,
3. Being admitted due to respiratory system disease,
4. Inhaler treatment with a nebulizer will be applied.

Exclusion Criteria:

1. Parent and child not voluntarily participating in the study,
2. Intravenous, intramuscular or any other treatment request,
3. The child has any genetic, congenital, chronic or metabolic disease,
4. The child has vision, hearing and speech problems,
5. The child's vital signs are unstable (no fever, tachypnea, etc.) and the need for any emergency intervention.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Reducing the child's fear | during inhaler treatment
  Reducing the child's fear during inhaler treatment
Reducing the child's anxiety | during inhaler treatment
  Reducing the child's anxiety during inhaler treatment

SECONDARY OUTCOMES:
Reducing the "Child Fear Scale" score | shortly after inhaler treatment
  The Child Fear Scale (CFS) used. This one-item scale consists of five sex-neutral faces. It ranges from a no fear (neutral) face on the far left to a face showing extreme fear on the far right. The rater responds indicates the level of fear. Scores range from 0 to 4.
Reducing the "Child Anxiety Scale-Stateness" score | shortly after inhaler treatment
  The Children's Anxiety Meter (CAM) used. It assesses children's anxiety in clinical settings and uses before medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom, also includes horizontal lines at intervals going up to the top. Children are asked to mark how he/she feel "right now" to measure state anxiety. Scores range from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No